CLINICAL TRIAL: NCT01174459
Title: Survey on Long-Term Use of BI-Sifrol® Tablets in Patients With Restless Legs Syndrome
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.678
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patient with Restless Legs Syndrome

SUMMARY:
The survey is conducted to investigate the safety and efficacy of long-term use of BI-Sifrol Tablets in Restless Legs Syndrome (RLS) patients with or without renal dysfunction in routine medical practice.

ELIGIBILITY:
Inclusion criteria:

Patient with Restless Legs Syndrome

Exclusion criteria:

None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 500
Sampling Method: Non-Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (159):
- Japan (159):
  - Boehringer Ingelheim Investigational Site 119, Akashi
  - Boehringer Ingelheim Investigational Site 52, Akishima
  - Boehringer Ingelheim Investigational Site 16, Akita
  - Boehringer Ingelheim Investigational Site 22, Ami-machi
  - Boehringer Ingelheim Investigational Site 36, Asahi
  - Boehringer Ingelheim Investigational Site 1, Asahikawa
  - Boehringer Ingelheim Investigational Site 40, Chiba
  - Boehringer Ingelheim Investigational Site 158, Chōfu
  - Boehringer Ingelheim Investigational Site 78, Chūō
  - Boehringer Ingelheim Investigational Site 66, Fujisawa
  - Boehringer Ingelheim Investigational Site 7, Fukagawa
  - Boehringer Ingelheim Investigational Site 144, Fukuoka
  - Boehringer Ingelheim Investigational Site 146, Fukuoka
  - Boehringer Ingelheim Investigational Site 19, Fukushima
  - Boehringer Ingelheim Investigational Site 132, Fukuyama
  - Boehringer Ingelheim Investigational Site 82, Gifu
  - Boehringer Ingelheim Investigational Site 83, Hamamatsu
  - Boehringer Ingelheim Investigational Site 56, Hatchioji
  - Boehringer Ingelheim Investigational Site 129, Hayashima-machi
  - Boehringer Ingelheim Investigational Site 123, Himeji
  - Boehringer Ingelheim Investigational Site 111, Hirakata
  - Boehringer Ingelheim Investigational Site 133, Hiroshima
  - Boehringer Ingelheim Investigational Site 30, Honjō
  - Boehringer Ingelheim Investigational Site 38, Ichihara
  - Boehringer Ingelheim Investigational Site 37, Ichikawa
  - Boehringer Ingelheim Investigational Site 79, Ichikawasango-machi
  - Boehringer Ingelheim Investigational Site 117, Ikeda
  - Boehringer Ingelheim Investigational Site 149, Isahaya
  - Boehringer Ingelheim Investigational Site 118, Itami
  - Boehringer Ingelheim Investigational Site 10, Iwamizawa
  - Boehringer Ingelheim Investigational Site 127, Izumo
  - Boehringer Ingelheim Investigational Site 154, Kagoshima
  - Boehringer Ingelheim Investigational Site 155, Kagoshima
  - Boehringer Ingelheim Investigational Site 74, Kanazawa
  - Boehringer Ingelheim Investigational Site 76, Kanazawa
  - Boehringer Ingelheim Investigational Site 120, Katō
  - Boehringer Ingelheim Investigational Site 124, Kawai-machi
  - Boehringer Ingelheim Investigational Site 60, Kawasaki
  - Boehringer Ingelheim Investigational Site 63, Kawasaki
  - Boehringer Ingelheim Investigational Site 31, Keroyama-machi
  - Boehringer Ingelheim Investigational Site 145, Kitakyuushu
  - Boehringer Ingelheim Investigational Site 122, Kobe
  - Boehringer Ingelheim Investigational Site 46, Kodaira
  - Boehringer Ingelheim Investigational Site 50, Kodaira
  - Boehringer Ingelheim Investigational Site 32, Koshigaya
  - Boehringer Ingelheim Investigational Site 101, Kōtari
  - Boehringer Ingelheim Investigational Site 150, Kumamoto
  - Boehringer Ingelheim Investigational Site 151, Kumamoto
  - Boehringer Ingelheim Investigational Site 143, Kurume
  - Boehringer Ingelheim Investigational Site 102, Kyoto
  - Boehringer Ingelheim Investigational Site 103, Kyoto
  - Boehringer Ingelheim Investigational Site 98, Kyoto
  - Boehringer Ingelheim Investigational Site 99, Kyoto
  - Boehringer Ingelheim Investigational Site 100, Maizuru
  - Boehringer Ingelheim Investigational Site 80, Matsumoto
  - Boehringer Ingelheim Investigational Site 81, Matsumoto
  - Boehringer Ingelheim Investigational Site 142, Matsuyama
  - Boehringer Ingelheim Investigational Site 28, Mibu-machi
  - Boehringer Ingelheim Investigational Site 138, Miki-machi
  - Boehringer Ingelheim Investigational Site 115, Minoo
  - Boehringer Ingelheim Investigational Site 47, Mitaka
  - Boehringer Ingelheim Investigational Site 153, Miyazaki
  - Boehringer Ingelheim Investigational Site 134, Miyoshi
  - Boehringer Ingelheim Investigational Site 112, Moriguchi
  - Boehringer Ingelheim Investigational Site 13, Morioka
  - Boehringer Ingelheim Investigational Site 2, Muroran
  - Boehringer Ingelheim Investigational Site 88, Nagakute-machi
  - Boehringer Ingelheim Investigational Site 41, Nagareyama
  - Boehringer Ingelheim Investigational Site 148, Nagasaki
  - Boehringer Ingelheim Investigational Site 85, Nagoya
  - Boehringer Ingelheim Investigational Site 86, Nagoya
  - Boehringer Ingelheim Investigational Site 87, Nagoya
  - Boehringer Ingelheim Investigational Site 92, Nagoya
  - Boehringer Ingelheim Investigational Site 68, Nigata-honmachi
  - Boehringer Ingelheim Investigational Site 69, Nigata-honmachi
  - Boehringer Ingelheim Investigational Site 70, Nigata-honmachi
  - Boehringer Ingelheim Investigational Site 71, Nigata-honmachi
  - Boehringer Ingelheim Investigational Site 139, Niihama
  - Boehringer Ingelheim Investigational Site 141, Niihama
  - Boehringer Ingelheim Investigational Site 11, Ninohe
  - Boehringer Ingelheim Investigational Site 121, Nishinomiya
  - Boehringer Ingelheim Investigational Site 157, Nishitōkyō
  - Boehringer Ingelheim Investigational Site 130, Okayama
  - Boehringer Ingelheim Investigational Site 131, Okayama
  - Boehringer Ingelheim Investigational Site 89, Okazaki
  - Boehringer Ingelheim Investigational Site 104, Osaka
  - Boehringer Ingelheim Investigational Site 105, Osaka
  - Boehringer Ingelheim Investigational Site 106, Osaka
  - Boehringer Ingelheim Investigational Site 17, Ōdate
  - Boehringer Ingelheim Investigational Site 152, Ōita
  - Boehringer Ingelheim Investigational Site 128, Ōta-ku
  - Boehringer Ingelheim Investigational Site 97, Ōtsu
  - Boehringer Ingelheim Investigational Site 140, Ōzu
  - Boehringer Ingelheim Investigational Site 26, Ryūgasaki
  - Boehringer Ingelheim Investigational Site 147, Saga
  - Boehringer Ingelheim Investigational Site 64, Sagamihara
  - Boehringer Ingelheim Investigational Site 34, Saitama
  - Boehringer Ingelheim Investigational Site 107, Sakai
  - Boehringer Ingelheim Investigational Site 108, Sakai
  - Boehringer Ingelheim Investigational Site 39, Sakura
  - Boehringer Ingelheim Investigational Site 3, Sapporo
  - Boehringer Ingelheim Investigational Site 4, Sapporo
  - Boehringer Ingelheim Investigational Site 5, Sapporo
  - Boehringer Ingelheim Investigational Site 6, Sapporo
  - Boehringer Ingelheim Investigational Site 8, Sapporo
  - Boehringer Ingelheim Investigational Site 9, Sapporo
  - Boehringer Ingelheim Investigational Site 113, Sayama
  - Boehringer Ingelheim Investigational Site 14, Sendai
  - Boehringer Ingelheim Investigational Site 15, Sendai
  - Boehringer Ingelheim Investigational Site 27, Shimotsuke
  - Boehringer Ingelheim Investigational Site 29, Shimotsuke
  - Boehringer Ingelheim Investigational Site 125, Shingū
  - Boehringer Ingelheim Investigational Site 84, Shizuoka
  - Boehringer Ingelheim Investigational Site 95, Suzuka
  - Boehringer Ingelheim Investigational Site 96, Suzuka
  - Boehringer Ingelheim Investigational Site 137, Takamatsu
  - Boehringer Ingelheim Investigational Site 109, Takatsuki
  - Boehringer Ingelheim Investigational Site 110, Takatsuki
  - Boehringer Ingelheim Investigational Site 12, Takizawa-mura
  - Boehringer Ingelheim Investigational Site 33, Tokorozawa
  - Boehringer Ingelheim Investigational Site 42, Tokyo Arakawa
  - Boehringer Ingelheim Investigational Site 53, Tokyo Chuo
  - Boehringer Ingelheim Investigational Site 43, Tokyo Itabashi
  - Boehringer Ingelheim Investigational Site 45, Tokyo Meguro
  - Boehringer Ingelheim Investigational Site 54, Tokyo Minato
  - Boehringer Ingelheim Investigational Site 49, Tokyo Nerima
  - Boehringer Ingelheim Investigational Site 55, Tokyo Nerima
  - Boehringer Ingelheim Investigational Site 44, Tokyo Ota
  - Boehringer Ingelheim Investigational Site 51, Tokyo Shibuya
  - Boehringer Ingelheim Investigational Site 58, Tokyo Shibuya
  - Boehringer Ingelheim Investigational Site 57, Tokyo Shinagawa
  - Boehringer Ingelheim Investigational Site 48, Tokyo Shinjyuku
  - Boehringer Ingelheim Investigational Site 21, Toride
  - Boehringer Ingelheim Investigational Site 126, Tottori
  - Boehringer Ingelheim Investigational Site 72, Toyama
  - Boehringer Ingelheim Investigational Site 73, Toyama
  - Boehringer Ingelheim Investigational Site 90, Toyohashi
  - Boehringer Ingelheim Investigational Site 93, Toyohashi
  - Boehringer Ingelheim Investigational Site 91, Toyokawa
  - Boehringer Ingelheim Investigational Site 94, Toyokawa
  - Boehringer Ingelheim Investigational Site 114, Toyonaka
  - Boehringer Ingelheim Investigational Site 116, Toyonaka
  - Boehringer Ingelheim Investigational Site 20, Tsuchiura
  - Boehringer Ingelheim Investigational Site 24, Tsukuba
  - Boehringer Ingelheim Investigational Site 77, Tsuruga
  - Boehringer Ingelheim Investigational Site 35, Tsurugashima
  - Boehringer Ingelheim Investigational Site 156, Urazoe
  - Boehringer Ingelheim Investigational Site 23, Ushiku
  - Boehringer Ingelheim Investigational Site 25, Ushiku
  - Boehringer Ingelheim Investigational Site 75, Utinada-machi
  - Boehringer Ingelheim Investigational Site 18, Yamagata
  - Boehringer Ingelheim Investigational Site 135, Yanai
  - Boehringer Ingelheim Investigational Site 59, Yokohama
  - Boehringer Ingelheim Investigational Site 61, Yokohama
  - Boehringer Ingelheim Investigational Site 62, Yokohama
  - Boehringer Ingelheim Investigational Site 65, Yokohama
  - Boehringer Ingelheim Investigational Site 67, Yokohama
  - Boehringer Ingelheim Investigational Site 159, Yokose-machi
  - Boehringer Ingelheim Investigational Site 136, Yoshinogawa

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient With Restless Legs Syndrome: Pramipexole immediate release tablets, oral administration, 0.125 mg/day to maximum 0.75 mg/day
Period: Overall Study
Arm/Group | Patient With Restless Legs Syndrome
Started | 571 (Registered patients)
Completed | 566 (Case report form (CRF) collected)
Not Completed | 5
Not completed — case report form (CRF) not collected | 5

BASELINE CHARACTERISTICS:
Population: Safety set: all patients who were documented to have taken at least one dose of pramipexole except for patients who had no observation documented after entry, made invalid registration or were not under the appropriate site contact.
  56 patients who didn't visit hospital after the treatment of pramipexole for RLS were excluded from safety set.
Arm/Group | Patient With Restless Legs Syndrome
Number analyzed (Participants) | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298
  Male | 212

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Drug-related Adverse Events
Description: Number of patients with drug-related adverse events
Time Frame: 12 Months
Population: Safety set: all patients who were documented to have taken at least one dose of pramipexole except for patients who had no observation documented after entry, made invalid registration or were not under the appropriate site contact.
Measure: Number; unit: participants
Arm/Group | Patient With Restless Legs Syndrome
Number analyzed (Participants) | 510
participants | 76

2. Secondary Outcome: Change From Baseline in Total Score of the International Restless Legs Syndrome Rating Scale (IRLS)
Description: International Restless Legs Syndrome rating scale (IRLS): The IRLS rating scale is a selfrating scale used to evaluate the severity of RLS and the patients are requested to answer 10 questions on a scale of 0 to 4. Respective scores (0-4 points) for the 10 questions were added up to calculate the total score on the IRLS. Therefore the total score is 0-40. The lower values represent a better outcome.
Time Frame: after 12 months or at the end of observation
Population: Efficacy set: The patient set included all patients in the safety set with approved indication RLS and had IRLS total score measurement at baseline and at least one post-baseline time point.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Patient With Restless Legs Syndrome
Number analyzed (Participants) | 407
Score on a scale | -13.42 (10.40)

ADVERSE EVENTS:
Time Frame: During the 12-month period or within 2 days after the last administration of pramipexole, up to 990 days.
Description: Number of participants at risk is based on safety set.
Arm/Group | Patient With Restless Legs Syndrome
Serious Adverse Events (participants affected / at risk) | 10/510
Other Adverse Events (participants affected / at risk) | 0/510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient With Restless Legs Syndrome (N=510)
Supraventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Impulse-control disorder (Psychiatric disorders) | 1
Somatic hallucination (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.